CLINICAL TRIAL: NCT03958721
Title: Concurrent Capecitabine and Radiotherapy in the Adjuvant Treatment of Resistant Breast Cancer: A Prospective Feasibility Trial
Brief Title: Capecitabine and Radiotherapy in the Adjuvant Treatment of Resistant Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: A Bapsi Chakravarthy, MD (Other)
Responsible Party: Sponsor-Investigator, A Bapsi Chakravarthy, MD, Professor; Radiation Oncology, Vanderbilt-Ingram Cancer Center
Organization: Vanderbilt-Ingram Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VICC BREP 1898; NCI-2019-03276 (Registry Identifier: NCI, Clinical Trials Reporting Program)
Record Dates: First submitted 2019-05-17; First posted 2019-05-22 (Actual); Last update posted 2023-11-27 (Actual); Status verified 2023-11

CONDITIONS: Resistant Breast Cancer; Non-metastatic Invasive Breast Cancer
MeSH Terms: interventions — Capecitabine; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Concurrent Adjuvant Capecitabine and Radiotherapy (Experimental)
  Interventions: Drug: Capecitabine; Radiation: Radiotherapy

INTERVENTIONS:
Drug: Capecitabine — 1,000 mg/m2 twice daily taken by mouth every other week
Radiation: Radiotherapy — Once daily (Monday through Friday) for six weeks

SUMMARY:
This is a single-arm, prospective, non-randomized, feasibility study evaluating concurrent capecitabine-radiotherapy in participants with Resistant Breast Cancer.

DETAILED DESCRIPTION:
Primary Objective:

- To evaluate the feasibility of a novel concurrent capecitabine-radiotherapy regimen by characterizing the percentage of patients who complete concurrent capecitabine-radiotherapy as a preliminary study before a larger trial.

Secondary Objectives

* To report the tolerability of concurrent capecitabine-radiotherapy with patient-reported HRQOL outcomes via RAND 36-Item Health Survey.
* To characterize radiation dermatitis secondary to concurrent capecitabine-radiotherapy through patient-reported RISR scores and to compare concurrent RISR scores to published reports of patients undergoing breast cancer radiotherapy only.
* To provide a preliminary description of the toxicity profile of concurrent capecitabine radiotherapy and report the frequency of grade 3 or grade 4 toxicity during combined therapy.
* To report the feasibility of completion of all study assessments, and completion of all study and exploratory assessments.

Outline:

This trial will investigate chemoradiotherapy with capecitabine at 1000 mg/m2 BID every other week during radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed non-metastatic invasive breast cancer who will be undergoing neoadjuvant chemotherapy and have persistent disease at time of definitive surgery

  * Tumors must have ER/PR/HER2 status reported by available pathology report(s)
  * Both triple negative and hormone receptor positive patients are eligible for enrollment
* Completion of neoadjuvant chemotherapy

  * May not include capecitabine or 5-FU containing regimens
  * Resolution of adverse events from neoadjuvant chemotherapy including biochemical/hematologic to CTCAE v5.0 grade 1 or below (except alopecia) prior to initiation of study therapy
  * Recovery time between surgery and study therapy ≥ 4 weeks.
* Persistent invasive disease following neoadjuvant chemotherapy in either the breast, lymph node, or both ). Any residual tumor; lack of complete pathologic response.
* Patients planning to receive adjuvant radiation to the breast and/or regional nodes.
* Patients planning to receive capecitabine per the treating physician

Patients already receiving capecitabine as adjuvant therapy are eligible to enroll in this study, provided adverse events deemed by the treating physician as possibly, probably or definitely related to adjuvant capecitabine prior to study therapy have resolved to CTCAE v.5.0 grade 1 or below (except alopecia), and provided duration of planned capecitabine includes entire duration of planned radiotherapy.

* ECOG performance status 0 or 1
* Tamoxifen: patients who have received Tamoxifen as chemoprevention are still eligible.

Endocrine receptor therapies (Hormone receptor inhibitors) may not be given with study treatment.

* . Patients who have had radiation to the contralateral breast are eligible.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Pregnant or lactating females. Women who are pregnant or who become pregnant are excluded from this study because capecitabine is a chemotherapeutic agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with capecitabine, breastfeeding should be discontinued if the mother is treated with capecitabine. These potential risks may also apply to radiotherapy used in this study.
* Serious medical or psychiatric illness that in the judgement of the treating physician places the patient at risk & would limit compliance with the study requirements.
* Inability to swallow or retain whole pills.
* Patients with known or suspected allergy to capecitabine or 5-FU.
* Contraindications to capecitabine or radiotherapy as determined by the treating physician including severe renal impairment (GFR < 30).
* Prior radiation to the ipsilateral breast.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 20 (Actual)
Dates: Start 2019-07-18 (Actual); Primary Completion 2023-10-26 (Actual); Study Completion 2023-10-26 (Actual)

PRIMARY OUTCOMES:
Percentage of patients who complete concurrent capecitabine-radiotherapy | Up to 6 months

SECONDARY OUTCOMES:
Assess tolerability | Up to 6 months
  Patient reported health-related quality of life outcomes via RAND 36-Item Health Survey HRQOL outcomes via RAND 36-Item Health Survey
Characterize radiation dermatitis secondary to concurrent capecitabine-radiotherapy | Up to 7 months
  Through patient-reported RISR scores
Frequency of grade 3-4 adverse events | Up to 7 months
  Events will be graded according to the National Cancer Institute Common Terminology
Completion of study study assessments | Up to 7 months
  Median number of study assessments completed
Completion of exploratory assessments | Up to 7 months
  Median number of exploratory assessment completed

CONTACTS AND LOCATIONS:
Overall Officials: Bapsi Chakravarthy, MD, Principal Investigator — Vanderbilt Medical Center
Locations (1):
- Vanderbilt-Ingram Cancer Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2022-02-02): https://cdn.clinicaltrials.gov/large-docs/21/NCT03958721/ICF_000.pdf